CLINICAL TRIAL: NCT02900339
Title: MRI Sequences Optimization in Healthy Subjects
Brief Title: Magnetic Resonance Imaging (MRI) Sequences Optimization in Healthy Subjects
Acronym: OSS-IRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC11_8965; 2011-A01531-40 (Other: Id-RCB)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers
Keywords: MRI; Sequence optimization; Healthy volunteers
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MR parameters optimization (Experimental): The study will be conducted on the MRI of the Neurinfo platform, in the radiology department of the University Hospital of Rennes.
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — MRI of the Neurinfo platform is an MRI 3 Tesla Magnetom Verio model, Siemens (Siemens Healthcare, Erlangen, Germany). This imager is marked for European Conformity (CE), ensuring compliance with European Union safety standards.
  Other Names: Magnetom

SUMMARY:
Magnetic resonance imaging (MRI) is a noninvasive and non-ionizing (no use of X-rays) imaging modality. Today it is considered an anatomical and functional exploration reference technique. Since its inception around 1985, this technology is constantly evolving.

Many advances in MRI require constant adaptations of radiological practices. The morphological image is now associated with functional and parametric information (infusion, diffusion spectroscopy, etc ...). In parallel, work combining acquisition and post-processing of data also open new applications (tractography, functional MRI, etc ....). Thus, more and more procedures are necessary to "integrate" these techniques for the diagnosis and adapt to new demands of clinicians.

The type of sequence and its associated parameters allow to directly influence the contrast of images, to characterize tissue compared to another and, ultimately, to highlight morphological or functional abnormality. Image quality can be optimized on each MRI, depending on the time available for the acquisition on the one hand, and on the desired resolution and contrast, on the other hand. For each sequence, it is therefore necessary to find a compromise that will optimize the diagnostic quality of the examination.

This optimization requires a phase focusing on healthy volunteers. It is therefore important that researchers and physicists could design on healthy volunteers, the best settings of all parameters for an image or spectrum. Indeed, it is always necessary to properly optimize every parameter choices before beginning a study of a cohort of patients.

In this context, the main objective of this study is to optimize sequences and imaging protocols to evaluate and validate the choice of parameters in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged over 18 years
* Written informed consent given

Exclusion Criteria:

* contraindication to MRI :

  * Claustrophobia
  * morphotype not allowing access to MRI
  * Wear a metallic implant, such as:
  * Pacemaker (pacemaker)
  * Ferromagnetic surgical clips
  * Intra orbital metallic foreign bodies or encephalic
* Pregnancy
* Breastfeeding
* Adults under guardianship, trusteeship or safeguard justice
* No social Insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2013-04-18 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Quantitative assessment of acquired sequences | One day after data acquisitions
  Quality images, maps or spectra acquired with optimized parameters will be compared to standard acquisitions.
  This evaluation will be based on quantitative criteria extracted from computer analysis of the data : signal to noise ratio, contrast-to-noise, blur level, information sharing, collocation of areas set evidenced by the different techniques, etc...

SECONDARY OUTCOMES:
Qualitative assessment of acquired sequences | One day after data acquisitions
  Quality images, maps or spectra acquired with optimized parameters will be compared to standard acquisitions.
  This evaluation will be based on statistical comparison of visual qualitative criteria by experts radiologists

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe FERRE, MD, PhD, Study Director — CHU Rennes
Locations (1):
- Radiology Department CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No